CLINICAL TRIAL: NCT01322412
Title: Adapted Physical Activity Effect on Aerobic Function and Fatigue in Patients With Breast Cancer Treated in Adjuvant Phase
Brief Title: Adapted Physical Activity Effect and Fatigue in Patients With Breast Cancer
Acronym: SAPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I10 009 / SAPA
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2011-03

CONDITIONS: Breast Cancer
Keywords: Adapted physical activity; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm A : physical activity program: Arm A : physical activity program (aerobic and strength training) during the 27 weeks of treatment (chemotherapy and radiotherapy) and conventional follow-up during 27 weeks
- Arm B : conventional management: Arm B : conventional management during and after treatment

SUMMARY:
Physical exercise has been identified as a major item of many chronic diseases and cancer rehabilitation.

Therefore, physical activity for health is a valid and relevant way to improve quality of life and to manage cancer patient fatigue. The aim of the study is the assessment of the effects of a physical activity retraining program on aerobic capacity, strength and fatigue, in a breast cancer population treated by adjuvant chemotherapy.

DETAILED DESCRIPTION:
Physical exercise has been identified as a major item of many chronic diseases and cancer rehabilitation. It contributes to an improvement in the quality of life and to a decrease in the current treatment side effects and mortality. Cancer in association with treatment toxicity and an inactive lifestyle lead to a fall in physical capability and causes problems in daily activities. The physical capacity and the tolerance for exercise fall simultaneously leading to a deconditioning vicious circle which increases physical, psychological and emotional symptoms of fatigue. Therefore, physical activity for health is a valid and relevant way to improve quality of life and to manage cancer patient fatigue. The aim of the study is the assessment of the effects of a physical activity retraining program on aerobic capacity, strength and fatigue, in a breast cancer population treated by adjuvant chemotherapy.

A total of 44 subjects is required. The programme is organised as follows: Arm A (aerobic and strength training) and during the 27 weeks of treatment (chemotherapy and radiotherapy); Arm B (control group). This study includes 3 assessments phases (T0: before adjuvant chemotherapy; T1 (week 27) and T2: final evaluation at the 54th week). These assessments include: cardiopulmonary exercise test including maximal oxygen uptake test (VO2max), six-minute walk test, muscular testing, assessment of physical activity (IPAQ questionnaire), fatigue (MFI20 questionnaire), quality of life (EORTC QLQ C30), anxiety and depression symptoms (HADS) and nutritional evaluation: BMI and total body photonic absorption.

ELIGIBILITY:
Inclusion Criteria:

* females between 18 and 75 years of age
* signed written informed consent
* willing to take part in the trial and to follow the instructions
* breast tumour, histologically documented
* patients who have undergone curative surgery
* patients for whom a 6-treatment course of adjuvant chemotherapy (3FEC100 + taxanes) and radiotherapy has been scheduled
* patients with HER2-negative cancer.

Exclusion Criteria:

* metastatic cancer
* other primary tumours
* disability preventing a proper understanding of the instructions for the trial
* chemotherapy strictly contra-indicated
* patients who are subject to a court protection, wardship or guardianship order
* uncontrolled hypertension
* family history of sudden death in a first-degree relative
* unstabilised heart disease
* current treatment with beta-blockers
* chronic or acute pulmonary disease associated with dyspnoea upon moderate effort
* uncontrolled thyroid dysfunction
* uncontrolled diabetes
* any other serious conditions that are unstabilised, disabling or in which physical exercise is contra-indicated
* unable to attend for follow-up throughout the duration of the study
* ventricular ejection fraction (vef) < 50%, pregnancy or suckling.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adjuvant breast cancer
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
main criterion is exercise tolerance at 27 weeks, measured by VO2 max, following a physical activity (PA) programme | 27 weeks

SECONDARY OUTCOMES:
Assessment at 27 and 54 weeks between the 2 groups of muscle function. | 54 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vincent FRANCOIS, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Limoges University Hospital, Limoges, France

REFERENCES:
- [Result] Cornette T, Vincent F, Mandigout S, Antonini MT, Leobon S, Labrunie A, Venat L, Lavau-Denes S, Tubiana-Mathieu N. Effects of home-based exercise training on VO2 in breast cancer patients under adjuvant or neoadjuvant chemotherapy (SAPA): a randomized controlled trial. Eur J Phys Rehabil Med. 2016 Apr;52(2):223-32. Epub 2015 May 19. PMID 25986222